CLINICAL TRIAL: NCT06564740
Title: Umbilical Cord Derived Mesenchymal Stem Cell (UC-MSC) Transplantation in Infants with Biliary Atresia: a Prospective Randomized Controlled Trial
Brief Title: Stem Cell Applications in Biliary Atresia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmi Kadıoğlu Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Azizoğlu, Medical Doctor, Necmi Kadıoğlu Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biliar Atresia Stem Cell
Record Dates: First submitted 2024-08-17; First posted 2024-08-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Biliary Atresia; Fibrosis, Liver; Stem Cell
Keywords: biliary atresia; liver fibrosis; stem cell
MeSH Terms: conditions — Biliary Atresia; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: This study is designed as a multicentric randomized controlled trial (RCT). Patients will be randomly divided into two groups. Treatment Group: 30 Kasai-operated BA patients who will receive UC-MSC transplantation, and Control Group: 30 BA patients who will only undergo Kasai operation. UC-MSC transplantation will be administered twice to each patient in the study group via the hepatic artery: the first transplantation will be performed post-surgery at the beginning, and the second one will be performed 6 months later, with a dose of 1 million UC-MSC/kg.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stem Cell Application Group (Experimental): In this group, UC-MSC transplantation will be administered twice to each patient in the study group via the hepatic artery: the first transplantation will be performed post-surgery at the beginning, and the second one will be performed 6 months later, with a dose of 1 million UC-MSC/kg. The applications will be applied after kasai portoenterostomy.
  Interventions: Drug: Stem Cell
- Control (Sham Comparator): In this group, UC-MSC will not be administered. This group serves as a passive control. The standard treatments that are routinely provided to Biliary Atresia patients will continue to be administered.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Stem Cell — UC-MSC transplantation will be administered twice to each patient in the study group via the hepatic artery: the first transplantation will be performed post-surgery at the beginning, and the second one will be performed 6 months later, with a dose of 1 million UC-MSC/kg.
  Arms: Stem Cell Application Group
Other: Control — In this group, UC-MSC will not be administered. This group serves as a passive control. The standard treatments that are routinely provided to these patients will continue to be administered.
  Arms: Control

SUMMARY:
Recently, mesenchymal stem cell (MSC) transplantation has emerged as a promising treatment for liver cirrhosis in adults. Additionally, bone marrow-derived stem cell transplantation has shown success in treating children with biliary atresia (BA). This study aims to evaluate the efficacy of Umbilical Cord-Derived Mesenchymal Stem Cell (UC-MSC) therapy in BA through a multicentric randomized controlled trial.

DETAILED DESCRIPTION:
Biliary atresia (BA) is the most common cause of chronic cholestasis in neonates and accounts for at least 50% of pediatric liver transplants. The incidence of BA is estimated to range from 1:5000 to 1:19000 live births. If the operation is not performed, all patients will die due to complications of liver cirrhosis. Recently, mesenchymal stem cell (MSC) transplantation has been found to be a promising treatment for liver cirrhosis in adults. Stem cell transplantation derived from bone marrow has also been successfully applied to children with BA. The aim of this study is to demonstrate the efficacy of Umbilical Cord-Derived Mesenchymal Stem Cell (UC-MSC) therapy in BA by planning a multicentric randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Infants were diagnosed with liver cirrhosis due to biliary atresia following Kasai's operation.
* The patients two months old or older and exhibited signs of cirrhosis after the procedure, including hepatomegaly, congestive splenomegaly, elevated liver enzymes, esophageal varices (confirmed by endoscopy), and cirrhosis (confirmed by liver biopsy).

Exclusion Criteria:

* Epilepsy
* Neurological disorders
* Coagulation disorders
* Diabetes
* Syndromic type biliary atresia
* Allergies to anesthetic agents
* Severe health conditions such as cancer or failure of the heart, lungs, liver, or kidneys, active infections, and severe psychiatric disorders.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 years
  Adverse events will be assessed during the stem cell applications, as well as at 1 week, 1 month, 3 months, 6 months, 1 year, and 2 years after the application.

SECONDARY OUTCOMES:
Pediatric End-Stage Liver Disease (PELD) score | 2 years
  Using PELD score (according to the suggestion of The Liver and Intestinal Organ Transplantation Committee in 2009). PELD is calculated based on three indicators: albumin (g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio). Formula: PELD = 10 * (0.48 * ln(Serum Bilirubin) + 1.857 * ln(INR) - 0.687 * ln(Albumin) + (0.436 if patient is less than 1 year old) + (0.667 if patient has growth failure)). Evaluate the result:
  If PELD <10: good results If 10 <PELD <15: average results If PELD> 15: bad results Albumin (Unit: g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio).
ALT levels (Alanine transaminase) | 2 years
  The levels of ALT will be closely monitored in both groups. The values for this parameter will be recorded and evaluated individually for each patient.
AST levels (Aspartate trasnaminase) | 2 years
  The levels of AST will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
Direct bilirubin levels | 2 years
  The levels of direct bilirubin will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
Total bilirubin levels | 2 years
  The levels of total bilirubin will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
GGT levels (Gama glutamil transferase) | 2 years
  The levels of GGT will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
Liver biopsy | 2 years
  Liver biopsy is a crucial clinical tool for assessing the progression and severity of cirrhosis
Level of cirrhosis | 2 years
  Level of cirrhosis will be assesed with PELD score. Using PELD score (according to the suggestion of The Liver and Intestinal Organ Transplantation Committee in 2009). PELD is calculated based on three indicators: albumin (g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio). Formula: PELD = 10 * (0.48 * ln(Serum Bilirubin) + 1.857 * ln(INR) - 0.687 * ln(Albumin) + (0.436 if patient is less than 1 year old) + (0.667 if patient has growth failure)). Evaluate the result:
  If PELD <10: good results If 10 <PELD <15: average results If PELD> 15: bad results Albumin (Unit: g / dL), bilirubin (units: mg / dL) and INR (international normalized ratio).
Re-operation rate | 2 years
  The patients who need further surgical intervention will be noted.
Liver transplantation | 2 years
  Liver transplantation will be evaluated. The number of patients requiring a liver transplant, along with the timing of the need, will be recorded.
Albumin levels | 2 years
  The levels of albumin will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
INR (international normalized ratio) | 2 years
  The levels of INR (international normalized ratio) will be closely monitored in both groups. The values for each parameter will be recorded and evaluated individually for each patient.
Cholangitis | 2 years
  The number of cholangitis for each cases will be closely monitored in both groups. The frequency of cholangitis experienced by each patient will be recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoglu, MD, PhD, Principal Investigator — Esenyurt State Hospital
Locations (1):
- Esenyurt State Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No